CLINICAL TRIAL: NCT05730504
Title: Evaluating the Effectiveness of a Mobile App-based Self-guided Psychological Interventions to Reduce Relapse in Substance Use Disorder: Protocol for a Randomized Controlled Trial
Brief Title: Evaluating the Effectiveness of Mobile Self-guided Psychological Interventions to Reduce Relapse in Substance Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PredictWatch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/003A
Record Dates: First submitted 2023-02-03; First posted 2023-02-15 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Substance Use Disorders; Addiction, Alcohol; Addiction, Substance
Keywords: mHealth; substance use disorder; alcohol; cannabis; stimulants
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app-based self-guided interventions (Experimental): Participants have access to self-guided, app-based mobile psychological interventions grounded in Cognitive Behavioral Therapy, meditation, mindfulness, journaling, as well as audio-guided sessions on gratitude, thoughts management, auto-empathy, and relaxation
  Interventions: Other: Mobile app-based self-guided interventions
- No interventions (No Intervention): Participants don't have access to app-based mobile psychological interventions

INTERVENTIONS:
Other: Mobile app-based self-guided interventions — self-guided, app-based mobile psychological interventions based on CBT, meditation, mindfulness, journaling, and audio-guided sessions on gratitude, thoughts management, auto-empathy, and relaxation
  Arms: Mobile app-based self-guided interventions

SUMMARY:
The aim of the study is to evaluate the effectiveness of mobile interventions in reducing craving and lapses in patients diagnosed with Substance Use Disorder. In a two-armed, randomized controlled trial the efficacy of self-guided psychological intervention delivered via a mobile app (Nałogometr 2.0) will be assessed. During the course of three months, participants will have access to intervention modules, based mainly on mindfulness and cognitive behavioral therapy (CBT). With the use of ecological momentary assessment (EMA), longitudinal data on several variables related to craving and lapse risk will be collected. Additionally, a questionnaire battery assessment - administered monthly - will measure severity of substance dependence, levels of anxiety, depression, and life satisfaction.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of mobile interventions in reducing craving and lapses in patients diagnosed with Substance Use Disorder.

Participants will be recruited from clinical patients receiving either in-patient or out-patient treatments for Substance Use Disorder (SUD) and enrolled in one of three groups: 1) Patients with alcohol addiction, 2) Patients with cross-addiction (alcohol and stimulants), 3) Patients with cannabis addiction.

Participants will be randomly assigned to either intervention or control condition. The mobile interventions will be delivered via a mobile app Nałogometr 2.0, freely available. Participants in the intervention condition will have free access to all of the app functionalities, while the control group won't gain access to the interventions until after study completion.

Interventions consist of audio-guided, short sessions on gratitude, thoughts management, motivation, relaxation, audio-guided mindfulness sessions concentrated on raising awareness of emotions and body signals or coping with stress, as well as CBT-based written sessions grounded in thought management and journaling techniques.

With the use of ecological momentary assessment (EMA), longitudinal data on several variables related to craving and lapse risk will be collected. Additionally, a questionnaire battery assessment - administered at baseline, after one month, after two months, and after three months - will measure severity of substance dependence, levels of anxiety, depression, and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a Substance Use Disorder (SUD)
* addiction to either alcohol, cannabis, or cross-addiction (alcohol + stimulants)
* min. 18 years of age
* fluent polish speakers
* users of Android or IOS smartphones

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
number of lapses | 3 months
  self-reported number of lapses collected during daily Ecological Momentary Assessment - an item asking if the lapse occurred since the last survey (yes / no). The frequency of lapses will be tracked for changes over time.
addiction craving | 3 months
  self-reported intensity of craving collected during daily Ecological Momentary Assessment - an item asking how strong is the urge to use on a scale from 0 to 6, where 0 means no urge, and 6 - an overwhelming urge. The score will be tracked for changes over time.

SECONDARY OUTCOMES:
Alcohol Use Disorder Identification Test (AUDIT) score | baseline, one month, two months, three months
  Problematic alcohol use will be measured with an Alcohol Use Disorders Identification Test (AUDIT). AUDIT assesses the amount and frequency of alcohol intake (items 1-3), alcohol dependence (questions 4-6), and problems related to alcohol consumption (items 7-10). Questions 1 to 8 are scored on a 5-point scale ranging from 0 to 4, and questions 9 and 10 are scored as 0, 2, or 4. Total scores range from 0 to 40, and the cut-off point to identify hazardous alcohol intake is 8, a score between 16 and 19 indicates harmful alcohol use, and scores above 20 points indicate possible alcohol use disorder. Participants will answer the questions in terms of standard drinks.
Severity of Dependence Scale (SDS) score | baseline, one month, two months, three months
  The Severity of Dependence Scale (SDS) will be used to provide a self-reported measure of psychological aspects of stimulants and alcohol dependence. A five-items, one-dimensional tool has uniform scale for questions 1 - 4 from 0 ('never or almost never') to 3 ('always'). Question 5 has the same scale with different signature where 0 means 'not difficult at all' and 3 means 'impossible'. Score ranging from 0 to 15, where cut-off score depends on user's drug type - a cut-off of =< 3 has been used for indexing alcohol dependence and =< 5 for indexing amphetamine dependence.
Cannabis Use Disorders Identification Test-Revised (CUDIT-R) score | baseline, one month, two months, three months
  Cannabis Use Disorders Identification Test-Revised (CUDIT-R) will be administered in a group of patients with cannabis addiction to assess cannabis consumption, abuse, dependence, and psychological features. The questionnaire consists of 7 items scored on a 0-4 scale, and the last question is scored on a three point scale (0-2-4). Scores of 8 or more indicate hazardous cannabis use, and the cut-off for possible cannabis use disorder is =<12 points.
Drug Use Disorders Identification Test (DUDIT) score | baseline, one month, two months, three months
  Drug Use Disorders Identification Test (DUDIT) is an 11-item screening questionnaire measuring drug intake and severity of substance ause and dependence. Items 1 to 9 are scored on a five-point Likert scale, and items 10 and 11 are scored on a three-point scale (0-2-4). Scores of 25 points or more are probably indicative of heavy dependence on drugs.
Hospital Depression and Anxiety Scale (HADS) score | baseline, one month, two months, three months
  Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with two subscales, each consisting of 7 items. For both subscales, scores between 8-10 indicate mild depression or anxiety, and scores in the range of 11-21 are indicative of depression or anxiety disorder.
Difficulties in Emotion Regulation Scale (DERS) score | baseline, one month, two months, three months
  Emotion regulation will be assessed with Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire, rated on a scale from 1 (almost never) to 5 (almost always). It consists of 6 subscales. Higher scores suggest greater difficulties in emotion regulation.
Satisfaction with Life Scale (SWLS) score | baseline, one month, two months, three months
  Participants' satisfaction with their life will be assessed with The Satisfaction With Life Scale (SWLS), Polish version from Jankowski (2015). SWLS is a short self-report instrument on which participants indicate their agreement to five statements about life satisfaction on a seven-point Likert scale. A maximum score of 35 can be reached, indicating a high level of life satisfaction.
Coping Orientation to Problems Experienced (mini-COPE) score | baseline, one month, two months, three months
  Coping Orientation to Problems Experienced (mini-COPE) questionnaire measures coping styles used to deal with difficult situations It consists of 28 items and three subscales corresponding to three coping styles. Higher scores on each of the subscale indicate increased usage of a corresponding coping style.
Impulsive Behavior Scale (SUPPS) score | baseline, one month, two months, three months
  Impulsive Behavior Scale (SUPPS) is a 20-item measure of impulsive traits. It consists of 20 items, with answers ranging from 1 = 'strongly agree' to 4 = 'strongly disagree'.
Brief Sensation Seeking Scale (BSSS) score | baseline, one month, two months, three months
  Brief Sensation Seeking Scale (BSSS) is a short, 8-item scale measuring sensation seeking. Responses are made on a 5-point scale, where higher score indicate stronger agreement. Higher scores indicate more impulsive behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- PredictWatch, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redel A, Binkowska AA, Obarska K, Marcowski P, Szymczak K, Lewczuk K, Solich K, Banaszak M, Woronowicz B, Nowicka M, Skorko M, Gola M, Bielecki M. Evaluating the effectiveness of a mobile app-based self-guided psychological interventions to reduce relapse in substance use disorder: protocol for a randomized controlled trial. Front Psychiatry. 2024 May 8;15:1335105. doi: 10.3389/fpsyt.2024.1335105. eCollection 2024. PMID 38784165